CLINICAL TRIAL: NCT04157803
Title: Accuracy of aCeTIC Acid to Predict Histopathology of Colonic Polyps
Acronym: Acetic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Aleman (Other)
Responsible Party: Principal Investigator, Federico Bentolila, Principal Investigator, Hospital Aleman
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HAleman
Record Dates: First submitted 2019-11-01; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient cohort (Other): Patients with polyps> 5mm with suspicion of tubular, tubulovillious or serrated adenomas, found during a videcolonoscopy.
  Interventions: Diagnostic Test: Acetic acid % spray

INTERVENTIONS:
Diagnostic Test: Acetic acid % spray — If during a videcolonoscopy a polyp is found with suspicion of tubular, tubulovillious or Serrated adenoma, the endoscopist will proceed to stain it using diffuser and acetic acid at a concentration of 3%. The presence or not of the aceto-whitening reaction will be evaluated, understanding it as the persistence of white staining of the polyp at one minute or three minutes, standing out from the surrounding mucosa.
  In case of positive staining it will be considered homogeneous if the staining is uniform on the surface of the polyp or heterogeneous if it is done irregularly.

SUMMARY:
The use of acetic acid in the characterization of polyps, produces a homogeneous white staining in sessile serrated adenomas, but not in tubular or tubulo-villous adenomas, a simple approach to predict polyp histopathology.

To determine the diagnostic accuracy of the use of acetic acid on tubular and serrated adenomas, during colonoscopy, a prospective diagnostic accuracy study was designed, taking as gold standard the pathological anatomy of the resected polyps.

Polyps found during a colonoscopy with suspicion of sessile serrated adenomas or tubular/tubulo villous will be included.

DETAILED DESCRIPTION:
In our experience tubular or tubulovillous adenomas with acetic acid have the same behavior as normal colonic mucosa. When sprayed with acetic acid they stain white, as well as the surrounding mucosa, but with a subsequent rapid loss of the effect. In contrast, serrated adenomas maintain an "aceto-whitening" reaction even though the surrounding normal mucosa loses staining.

The objectives are to determine the sensitivity and specificity, positive and negative probability coefficients of the positive or negative aceto-whitening reaction on serrated adenomas and tubular-tubulo-villous adenomas.

To determine the diagnostic accuracy of the use of acetic acid on tubular, tubulo-villous and serrated adenomas a prospective diagnostic accuracy study was designed considering the gold standard as the pathological anatomy of resected polyps.

As independent variables the presence or absence of aceto-whitening reaction after staining and the diagnostic impression of the endoscopist without acetic acid are considered. The presence or not of the aceto-whitening reaction will be evaluated, understanding it as the persistence of white staining of the polyp at one minute or three minutes, standing out from the surrounding mucosa.

In case of positive staining it will be considered homogeneous if the staining is uniform on the surface of the polyp or heterogeneous if it is done irregularly.

Place: German Hospital, endoscopy unit.

Data analysis: the data collected in double-entry tables will be captured to obtain the same sensitivity, specificity and positive or negative probability coefficients.

Sample size: 100 polyps.

Estimated duration: 1 month

ELIGIBILITY:
Inclusion Criteria:

* Patients with colonic polyps> 5mm with suspicion of tubular, tubulovillious or serrated adenomas, found during a videoolonoscopy.

Exclusion Criteria:

* Known acetic acid allergy
* Known or documented history of adenomatous or serrated polyposis
* Patients with inflammatory bowel disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-25 (Actual); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-11-15 (Estimated)

PRIMARY OUTCOMES:
Staining behaviour of the polyps after acetic acid: presence or absence of aceto-whitening reaction | 1 month
  The presence or not of the aceto-whitening reaction will be evaluated, understanding it as the persistence of white staining of the polyp at one minute or three minutes, standing out from the surrounding mucosa. In case of positive staining it will be considered homogeneous if the staining is uniform on the surface of the polyp or heterogeneous if it is done irregularly. This outcome will be evaluated visually by the involved endoscopist.
Histopathology of resected polyps | 1 month
  Histopathology of resected polyps defined by the observation of the resected specimen by a trained Pathologist.

SECONDARY OUTCOMES:
Histopathology impression of the endoscopist without acetic acid after resection. | 1 month
  Diagnostic guess of the endoscopist without acetic acid taking into account the shape of the polyp defined in the Paris classification and Kudo's pitt pattern

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Cimmino, MD, Principal Investigator — ENDIBA SAGE
Locations (1):
- Hospital Aleman, CABA, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Popoutchi P, Mota FL, Averbach M, de Menezes MS, Coudry RA. Acetic acid spray contribution in the endoscopic diagnosis of serrated polyposis syndrome. VideoGIE. 2018 Jan 5;3(2):65-67. doi: 10.1016/j.vgie.2017.11.011. eCollection 2018 Feb. No abstract available. PMID 29905183